CLINICAL TRIAL: NCT04574479
Title: Impact of Supra-inguinal Fascia Iliaca Compartment Block on Postoperative Opioid Consumption in Total Hip Arthroplasty Interventions by Posterior Approach
Brief Title: Supra-inguinal Fascia Iliaca Compartment Block on Postoperative Management in Total Hip Arthroplasty by Posterior Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Department, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/67
Record Dates: First submitted 2020-08-31; First posted 2020-10-05 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Arthropathy of Hip

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Two group simple-blinded RCT: placebo vs fascia iliaca group. Surgeon and patient are blinded of the patient's group. Investigator and loco-regional technique provider know the patient's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo group: patients have multimodal analgesia without fascia-iliaca compartment block
  Interventions: Drug: Multimodal analgesia and PCA morphine pump
- Fascia iliaca block (Experimental): Patients in this arm have multimodal analgesia with supra-inguinal fascia iliaca compartment block before surgery
  Interventions: Procedure: Supra-inguinal fascia iliaca compartment block; Drug: Multimodal analgesia and PCA morphine pump

INTERVENTIONS:
Procedure: Supra-inguinal fascia iliaca compartment block — Ultrasound guided loco-regional technique as described by Desmet et al. Fascia iliaca compartment block with in-plane 40 ml ropivacaine 0,375% injection between the ilio-psoas muscle and the internal oblique muscle.
  Patients in SFICB group have classical multimodal approach to postoperative analgesia with morphine administration by PCA pump
  Arms: Fascia iliaca block
Drug: Multimodal analgesia and PCA morphine pump — Patients in placebo group have classical multimodal approach to postoperative analgesia with morphine administration by PCA pump

SUMMARY:
Find the impact of supra-inguinal fascia iliaca compartment block on postoperative pain management after total hip arthroplasty by posterior surgical approach

DETAILED DESCRIPTION:
ASA physical status 1, 2 and 3 patients scheduled to undergo elective surgery of total hip arthroplasty under spinal anesthesia.

The investigators would like to study the impact of supra-inguinal fascia iliaca block on postoperative pain management after total hip arthroplasty by posterior surgical approach. The principal investigator perform this block with ultrasound technique. The investigators also want to observe if this loco-regional new approach to fascia iliaca block could have influence on opioid side effects, postoperative nausea and vomiting, length of hospitalisation and first mobilisation side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients scheduled to undergo elective surgery of total hip arthroplasty by posterior surgical aboard

Exclusion Criteria:

* Patient refusal
* Allergy to used medications or local infection.
* Pregnancy
* Obesity with body mass index > 35
* History of chronic pain or fibromyalgia
* Drug (opioids) addiction
* Treatment with corticosteroids for more than 6 months
* Severe kidney or liver diseases
* Mental disorders or serious neurological diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Opioid sparing | 48 hours after the intervention
  Difference in cumulated morphine consumption in the first 48 hours after surgery

SECONDARY OUTCOMES:
Opioid secondaries effects | 48 hours after the intervention
  incidence of secondary effects related to morphine consumption
Pain management satisfaction: questionnaire | 48 hours after the intervention
  pain management satisfaction score by IPO (International Pain Outcomes) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desmet M, Balocco AL, Van Belleghem V. Fascia iliaca compartment blocks: Different techniques and review of the literature. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):57-66. doi: 10.1016/j.bpa.2019.03.004. Epub 2019 Apr 17. PMID 31272654
- [Derived] Carella M, Beck F, Piette N, Denys S, Kurth W, Lecoq JP, Bonhomme VL. Effect of suprainguinal fascia iliaca compartment block on postoperative opioid consumption and functional recovery in posterolateral-approached total hip arthroplasty: a single-blind randomized controlled trial. Reg Anesth Pain Med. 2022 Jun 15:rapm-2021-103427. doi: 10.1136/rapm-2021-103427. Online ahead of print. PMID 35705263